CLINICAL TRIAL: NCT07351994
Title: Autonomic Neural Field Block for Visceral Pain Control in Minimally Invasive Left-Sided Colorectal Resections
Brief Title: Autonomic Neural Field Block for Visceral Pain in Minimally Invasive Left-Sided Colectomy
Acronym: ANfiELD
Status: Not yet recruiting | Type: Observational
Sponsor: Antonio Caycedo, MD (Other)
Responsible Party: Sponsor-Investigator, Antonio Caycedo, MD, Chief of Colorectal Surgery, Orlando Health, Inc.
Organization: Orlando Health, Inc. (Other)
Other Study IDs: 2365950-1
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain; Postoperative Nausea; Opioid Use
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Nerve Block

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Autonomic Neural Field Block Cohort: This cohort includes adult patients undergoing elective minimally invasive (laparoscopic or robotic) left-sided colonic or rectal resection with primary anastomosis who receive an intraoperative autonomic neural field block targeting the superior hypogastric and inferior mesenteric plexuses. The autonomic neural field block is performed under direct visualization as an adjunct to standard perioperative care within established enhanced recovery after surgery (ERAS) pathways. Use of additional analgesic modalities, including transversus abdominis plane blocks, non-opioid analgesics, and opioids, is permitted according to institutional practice and is recorded as part of routine perioperative management.
  Interventions: Procedure: Autonomic Neural Field Block

INTERVENTIONS:
Procedure: Autonomic Neural Field Block — An intraoperative autonomic neural field block targeting the superior hypogastric and inferior mesenteric plexuses is performed under direct visualization during elective minimally invasive left-sided colorectal resection. The block is administered using incremental injections of diluted local anesthetic as an adjunct to standard perioperative analgesic care within established enhanced recovery after surgery (ERAS) pathways.
  Other Names: Neural blockade

SUMMARY:
Effective postoperative pain control is a core component of enhanced recovery after surgery (ERAS) pathways in colorectal surgery; however, postoperative pain following minimally invasive left-sided colectomy remains a persistent clinical challenge. Standard multimodal analgesic strategies primarily target somatic pain pathways and may inadequately address visceral postoperative pain, which is mediated through autonomic afferent neural pathways. Residual visceral pain is associated with increased opioid consumption, postoperative nausea and vomiting, delayed recovery, and prolonged length of stay.

This prospective, multicenter observational registry evaluates the feasibility and real-world outcomes of an intraoperative autonomic neural field block targeting the superior hypogastric and inferior mesenteric plexuses during minimally invasive left-sided colectomy. The technique is performed under direct visualization as an adjunct to standard ERAS-based analgesic care. The primary outcome is postoperative opioid consumption within the first 24 hours after surgery. Secondary outcomes include opioid use through 48 hours, postoperative nausea and vomiting, antiemetic use, pain scores, length of stay, and readiness for discharge. Data from this registry will inform future comparative studies and help define the role of autonomic neural modulation in perioperative pain management for colorectal surgery.

DETAILED DESCRIPTION:
Background and Rationale

Effective postoperative pain control is a cornerstone of enhanced recovery after surgery (ERAS) pathways in colorectal surgery. Adequate analgesia facilitates early mobilization, pulmonary hygiene, gastrointestinal recovery, and timely hospital discharge. Despite widespread adoption of ERAS protocols and multimodal, opioid-sparing analgesic strategies, postoperative pain following left-sided colectomy remains a clinically relevant and persistent challenge. A substantial proportion of patients continue to experience moderate to severe pain in the early postoperative period, which may contribute to increased opioid consumption, postoperative nausea and vomiting (PONV), delayed functional recovery, and prolonged length of stay.

Current perioperative analgesic approaches in colorectal surgery predominantly address somatic pain pathways. These strategies include non-opioid analgesics, opioid-based regimens, local anesthetic infiltration, neuraxial techniques, and transversus abdominis plane (TAP) blocks. While effective in reducing abdominal wall and incisional pain, these modalities do not specifically target visceral postoperative pain, which is mediated through autonomic afferent neural pathways. Visceral pain arises from bowel distension, traction, ischemia, and inflammatory processes affecting the colon and mesentery and is transmitted primarily via sympathetic and parasympathetic fibers. This component of postoperative pain is qualitatively distinct, often diffuse and poorly localized, and frequently associated with nausea, ileus, and other autonomic symptoms.

Neuraxial techniques may provide effective visceral analgesia but are invasive, resource-intensive, and associated with potential adverse effects such as hypotension and urinary retention. As a result, many contemporary ERAS pathways have moved away from routine neuraxial analgesia, creating an unmet need for effective, targeted visceral pain control that is compatible with minimally invasive surgical workflows and ERAS principles.

Targeted modulation of autonomic neural pathways involved in visceral afferent transmission represents a potential strategy to address this gap. The superior hypogastric plexus and inferior mesenteric plexus play central roles in transmitting visceral sensory input from the left colon and rectum and are anatomically consistent structures routinely encountered during left-sided colorectal resection. Intraoperative autonomic neural field block targeting these plexuses may offer a mechanistically distinct approach to perioperative analgesia that complements existing somatic-focused techniques.

Description of the Intervention

The autonomic neural field block is performed intraoperatively during elective minimally invasive (laparoscopic or robotic) left-sided colonic or rectal resection with primary anastomosis constructed above the peritoneal reflection. Following establishment of pneumoperitoneum and trocar placement according to surgeon preference, standard minimally invasive dissection is carried out.

Dissection exposes the inferior mesenteric plexus in proximity to the origin of the inferior mesenteric artery and the superior hypogastric plexus at the level of the sacral promontory. These anatomic landmarks are routinely visualized during left-sided colorectal surgery and do not require additional dissection beyond standard operative technique.

An insulin needle connected to an anesthesia extension set is introduced through a 10-12 mm auxiliary port and attached to a syringe containing a diluted local anesthetic solution. All air is purged from the system prior to injection. Each plexus is infiltrated with approximately 5-7 mL of local anesthetic solution, administered incrementally in 1 mL aliquots. Aspiration is performed prior to each injection to confirm the absence of intravascular placement, and adequate tissue infiltration is confirmed visually. The surgical procedure then proceeds according to standard operative practice. When an extraction incision is used, any remaining local anesthetic solution may be infiltrated into the incision prior to closure.

Perioperative Analgesic Management

The autonomic neural field block is intended to complement, rather than replace, established multimodal perioperative analgesic strategies. Additional analgesic interventions, including TAP blocks, non-opioid medications, and opioid administration, are performed according to institutional ERAS protocols and surgeon or anesthesiologist discretion. This pragmatic approach allows evaluation of autonomic neural blockade within real-world clinical environments and across varying perioperative practices.

Study Design and Registry Framework

This study is a prospective, multicenter observational registry designed to systematically collect perioperative analgesic and recovery outcomes in patients undergoing minimally invasive left-sided colectomy who receive an intraoperative autonomic neural field block. The registry is descriptive and hypothesis-generating and does not mandate a comparator group. Use of additional analgesic modalities, including TAP block, is recorded but not standardized.

Participating centers collect perioperative data using standardized case report forms. Data capture includes patient demographics, operative details, analgesic interventions, and postoperative recovery metrics. The registry is designed to facilitate assessment of feasibility, reproducibility, and variability of outcomes across institutions and practice settings.

Outcome Measures

The primary outcome is postoperative opioid consumption, expressed as morphine milligram equivalents (MME), during the first 24 hours following surgery. Secondary outcomes include cumulative opioid consumption during the first 48 postoperative hours, intraoperative analgesic requirements, incidence of postoperative nausea and vomiting, antiemetic use, length of hospital stay, and readiness for discharge based on ERAS-aligned criteria. Patient-reported pain outcomes are collected during hospitalization and through the first postoperative week after discharge.

Safety and Feasibility

Feasibility outcomes include the ability to perform the autonomic neural field block under direct visualization without deviation from standard operative technique or prolongation of operative time. Adverse events potentially related to the intervention, including bleeding, vascular injury, or hemodynamic instability temporally associated with the block, are recorded. The registry does not alter routine postoperative monitoring or follow-up.

Data Analysis and Future Directions

Data from this registry will be summarized using descriptive statistics. The registry is not powered to assess comparative efficacy but is intended to generate preliminary data regarding analgesic patterns, recovery trajectories, and variability across centers. These findings will inform the design of future comparative or randomized studies, refine patient selection, and help define the role of autonomic neural modulation within ERAS-aligned perioperative pain management strategies for colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Scheduled for elective minimally invasive (laparoscopic or robotic) left-sided colonic or rectal resection with primary anastomosis constructed above the peritoneal reflection (e.g., sigmoid colectomy, left colectomy, anterior resection/rectosigmoid resection with intraperitoneal anastomosis).
* Planned intraoperative administration of autonomic neural field block targeting the superior hypogastric plexus and/or inferior mesenteric plexus, performed under direct visualization, as part of routine operative workflow.
* Managed perioperatively under an institutional standard analgesic pathway (e.g., ERAS or equivalent), with postoperative opioid administration recorded in the medical record.
* Ability to provide informed consent

Exclusion Criteria:

* Emergency/urgent colorectal surgery (e.g., perforation, uncontrolled bleeding, toxic megacolon, obstructing cancer requiring urgent operation).
* Planned open left-sided colectomy/rectal resection (minimally invasive approach not intended).
* Procedures in which no primary anastomosis is created (e.g., Hartmann's procedure, end colostomy, permanent diversion without anastomosis).
* Planned low pelvic/extra-peritoneal anastomosis (e.g., low anterior resection with anastomosis at or below the peritoneal reflection) or planned handsewn coloanal anastomosis.
* Known allergy or contraindication to the local anesthetic agents used for the block (or inability to receive local anesthetic for clinical reasons).
* Inability to reliably capture outcome data for the primary endpoint (e.g., anticipated transfer to another facility within 24 hours post-op, incomplete medication administration records).
* Pregnancy
* Prisoners or other protected populations where participation is restricted
* Chronic opioid therapy at baseline defined as daily opioid use for > 30 days preoperatively, or baseline opioid dose > 30 MME/day
* Planned use of neuraxial analgesia (epidural/spinal) intended for postoperative analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients undergoing elective minimally invasive (laparoscopic or robotic) left-sided colonic or rectal resection with primary anastomosis constructed above the peritoneal reflection. Eligible patients receive an intraoperative autonomic neural field block targeting the superior hypogastric and/or inferior mesenteric plexuses under direct visualization as part of routine operative care. Perioperative management follows institutional standardized analgesic pathways, such as enhanced recovery after surgery (ERAS) protocols, with postoperative opioid administration documented in the medical record. Patients undergoing emergency surgery, procedures without primary anastomosis, low pelvic or extraperitoneal anastomoses, planned open surgery, or those with contraindications to local anesthetics are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Opiod consumption | 24 hours
  Total opioid consumption during the first 24 hours following surgery, converted to morphine milligram equivalents (MME), based on all opioid medications administered during the postoperative period.

SECONDARY OUTCOMES:
Postoperative opioid consumption (48 hours) | 48 hours
  Total cumulative opioid consumption during the first 48 hours following surgery, converted to morphine milligram equivalents (MME), based on all opioid medications administered postoperatively
Intraoperative opioid administration | Intraoperative period
  Total opioid dose administered intraoperatively, converted to morphine milligram equivalents (MME), as recorded in the anesthesia record.
Postoperative nausea and vomiting (PONV) | First 48 hours after surgery
  Incidence of postoperative nausea and/or vomiting documented during the postoperative period and/or requirement for antiemetic medication.
Antiemetic medication use | First 48 hours after surgery
  Administration of any antiemetic medication during the postoperative period, recorded as a binary outcome and by total number of doses administered.
Postoperative pain intensity | Postoperative days 0-7
  Patient-reported pain intensity measured using a standardized numeric rating scale (0-10) at predefined postoperative time points.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Caycedo, MD, MSc, Principal Investigator — Orlando Health Colon & Rectal Institute

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: at 3,6 moths and after final results prior to any publication submission
Access Criteria: Reasonable request

REFERENCES:
- [Background] Daes J, Morrell DJ, Hanssen A, Caballero M, Luque E, Pantoja R, Luquetta J, Pauli EM. Paragastric Autonomic Neural Blockade to Prevent Early Visceral Pain and Associated Symptoms After Laparoscopic Sleeve Gastrectomy: a Randomized Clinical Trial. Obes Surg. 2022 Nov;32(11):3551-3560. doi: 10.1007/s11695-022-06257-9. Epub 2022 Sep 2. PMID 36050617
- [Result] Caycedo-Marulanda A, Sanchez A, Ferrara M, Daes J. Intraoperative autonomic field block combined with the transversus abdominis plane block: for left-sided colectomies (video forum). Tech Coloproctol. 2025 May 21;29(1):117. doi: 10.1007/s10151-025-03154-y. No abstract available. PMID 40397141